CLINICAL TRIAL: NCT01019629
Title: Expanded Screening for Fabry Trait
Brief Title: Fabry Screening Study
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 008-230
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Fabry Disease
Keywords: Fabry, Fabry Disease, Alpha-galactosidase A deficiency, GLA gene, mutations
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine if patients with a deficiency of alpha-galactosidase A are at-risk for cardiac complications that commonly occur in the general population

DETAILED DESCRIPTION:
Fabry disease is an X-linked deficiency of alpha-galactosidase A resulting primarily in an accumulation of globotriaosylceramide (Gb3) in virtually all organs and systems. The main complications of Fabry disease are a 20-fold increased risk of ischemic stroke, cardiac disease including cardiomyopathy, atrio-ventricular conduction defects, a wide variety of arrhythmias, valvular dysfunction (insufficiency or stenosis) and cardiac vascular disease as well as progressive renal failure. Fabry disease cannot be easily diagnosed in patients with routine EKGs, echocardiograms or MRIs. Screening non-selected at-risk populations of patients with ischemic stroke or cardiac disease for urinary Gb3, alpha-galactosidase A activity and GLA gene mutations should enable the identification of patients previously undiagnosed with Fabry disease among the general population of patients with heart disease and stroke

ELIGIBILITY:
Inclusion Criteria:

* Any diagnosis of heart disease.
* Male or Female
* Able to donate 12 cc of whole blood and 10 cc of urine

Exclusion Criteria:

* No diagnosis of cardiac disease.
* Unable to donate 12 cc of whole blood and/or 10 cc of urine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with any type of cardiac diagnosis
Sampling Method: Probability Sample
Enrollment: 2724 (Actual)
Dates: Start 2009-01-29 (Actual); Primary Completion 2013-04-17 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Identify GLA gene variants | Once
  Collect blood and urine sample one time only for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Schiffmann, M.D., M.H.Sc., Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor Institute of Metabolic Disease, Dallas, Texas, United States

REFERENCES:
- [Derived] Schiffmann R, Forni S, Swift C, Brignol N, Wu X, Lockhart DJ, Blankenship D, Wang X, Grayburn PA, Taylor MR, Lowes BD, Fuller M, Benjamin ER, Sweetman L. Risk of death in heart disease is associated with elevated urinary globotriaosylceramide. J Am Heart Assoc. 2014 Feb 4;3(1):e000394. doi: 10.1161/JAHA.113.000394. PMID 24496231